Effect of Monazite Sands in Patients with Osteoarthritis of the Knee Ethical committee Protocol No: 3.160.891

Pharmaceutical\_log

Documente date: May 3<sup>rd</sup> , 2019

## PHARMACEUTICAL LOG

**10.** At present, which drugs do you use that have been prescribed by your doctor? OBS: Observe the last prescriptions of the patient.

**Signature of the Principal Investigator:** 

| <b>Drug</b><br>( active principle and<br>trade name if any) | Brand<br>Generic<br>Similar | Posology | Who<br>prescribed¿ | Do you know<br>what you are<br>taking for this<br>medicine? If<br>yes, for what? | How do you<br>use this<br>medicine?<br>(See if use is<br>incorrect) | Since when<br>do you use<br>this<br>medication?<br>(days /<br>months /<br>years)) | After you started taking this medicine, did you feel any different reaction in the body? (any adverse reactions?) If yes, which one? | Did you get this medication at the SUS pharmacy or at a private pharmacy? Specify the location and how (free / paid) the patient purchased the medicine |
|---|---|---|---|---|---|---|---|---|
| 1 - | | | | | | | | |
| 2 - | | | | | | | | |
| 3 - | | | | | | | | |
| 4 - | | | | | | | | |
| 5 - | | | | | | | | |

Date:

| 11. What is your educational level? () DK / NR |
|---|
| 12. You could report your family income () Yes, what amount? () No () DK / NR |
| 13. How many people live with you? people |